CLINICAL TRIAL: NCT00536601
Title: Autologous Blood and Marrow Transplantation for Hematologic Malignancies and Selected Solid Tumors
Brief Title: High-Dose Chemotherapy With or Without Total-Body Irradiation Followed by Autologous Stem Cell Transplant in Treating Patients With Hematologic Cancer or Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 72806; NCI-2011-00131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 72806 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (PNET); Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Plasma Cell Neoplasm; Primary Systemic Amyloidosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Neuroblastoma; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Regional Neuroblastoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Neuroectodermal Tumors, Primitive, Peripheral; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Neuroblastoma; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Etoposide; Cyclophosphamide; Carmustine; Melphalan; Busulfan; Carboplatin; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Regimen CBV (patients with HL or NHL) (Experimental): Patients receive etoposide intravenously (IV) continuously over 34 hours on day -8, cyclophosphamide IV over 2 hours on days -7 to -4, and carmustine IV over 2 hours on day -3. Patients undergo ASCT on day 0.
  Interventions: Drug: etoposide; Drug: cyclophosphamide; Drug: carmustine; Procedure: autologous hematopoietic stem cell transplantation
- Regimen M200/M120 (patients with MM or amyloidosis) (Experimental): Patients receive 200 or 120 mg/m^2 of melphalan IV over 30 minutes on day -2. Patients undergo ASCT on day 0.
  Interventions: Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation
- Regimen BuC2iv (patients with ALL, AML, HL, or NHL) (Experimental): Patients receive busulfan IV over 2 hours then every 6 hours on days -7 to -4 for 16 total doses and cyclophosphamide IV over 2 hours on days -3 and -2. Patients undergo ASCT on day 0.
  Interventions: Drug: cyclophosphamide; Drug: busulfan; Procedure: autologous hematopoietic stem cell transplantation
- Regimen CT6 (patients with ALL) (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -5 to -4. Patients then undergo TBI twice daily on days -3 to -1. Patients undergo ASCT on day 0.
  Interventions: Drug: cyclophosphamide; Radiation: total-body irradiation; Procedure: autologous hematopoietic stem cell transplantation
- Regimen CTtCp (patients with other solid tumors) (Experimental): Patients receive cyclophosphamide IV continuously, carboplatin IV continuously, and thiotepa IV continuously over 24 hours on days -7 to -4. Patients undergo ASCT on day 0.
  Interventions: Drug: cyclophosphamide; Drug: carboplatin; Drug: thiotepa; Procedure: autologous hematopoietic stem cell transplantation
- Regimen VCp (patients with testicular cancer) (Experimental): Patients receive etoposide IV over 2-3 hours and carboplatin IV over 30 minutes on days -6 to -4. Patients undergo ASCT on day 0. At least 4 weeks after the first transplant, patients receive etoposide IV over 2-3 hours and carboplatin IV over 30 minutes on days -6 to -4. Patients then undergo a second ASCT on day 0.
  Interventions: Drug: etoposide; Drug: carboplatin; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation
- Regimen TtC1500/ECpM (patients with NBL or SRBCT) (Experimental): Patients receive thiotepa IV over 2 hours on days -7 to -5 and cyclophosphamide IV over 2 hours on days -5 to -2. Patients undergo ASCT on day 0. At least 4 weeks after the first transplant, patients receive carboplatin IV continuously over 24 hours on days -7 to -4, etoposide IV continuously over 24 hours on days -7 to -4, and melphalan IV over 30 minutes on days -7 to -5. Patients undergo a second ASCT on day 0.
  Interventions: Drug: etoposide; Drug: cyclophosphamide; Drug: melphalan; Drug: carboplatin; Drug: thiotepa; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Regimen CBV (patients with HL or NHL); Regimen TtC1500/ECpM (patients with NBL or SRBCT); Regimen VCp (patients with testicular cancer)
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Regimen BuC2iv (patients with ALL, AML, HL, or NHL); Regimen CBV (patients with HL or NHL); Regimen CT6 (patients with ALL); Regimen CTtCp (patients with other solid tumors); Regimen TtC1500/ECpM (patients with NBL or SRBCT)
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
  Arms: Regimen CBV (patients with HL or NHL)
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
  Arms: Regimen M200/M120 (patients with MM or amyloidosis); Regimen TtC1500/ECpM (patients with NBL or SRBCT)
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
  Arms: Regimen BuC2iv (patients with ALL, AML, HL, or NHL)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Regimen CTtCp (patients with other solid tumors); Regimen TtC1500/ECpM (patients with NBL or SRBCT); Regimen VCp (patients with testicular cancer)
Drug: thiotepa — Given IV
  Other Names: Oncotiotepa; STEPA; TESPA; Tespamin; TSPA
  Arms: Regimen CTtCp (patients with other solid tumors); Regimen TtC1500/ECpM (patients with NBL or SRBCT)
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
  Arms: Regimen CT6 (patients with ALL)
Procedure: autologous hematopoietic stem cell transplantation — Undergo ASCT
  Arms: Regimen BuC2iv (patients with ALL, AML, HL, or NHL); Regimen CBV (patients with HL or NHL); Regimen CT6 (patients with ALL); Regimen CTtCp (patients with other solid tumors); Regimen M200/M120 (patients with MM or amyloidosis)
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation — Undergo tandem ASCT
  Arms: Regimen TtC1500/ECpM (patients with NBL or SRBCT); Regimen VCp (patients with testicular cancer)

SUMMARY:
This pilot trial studies different high-dose chemotherapy regimens with or without total-body irradiation (TBI) to compare how well they work when given before autologous stem cell transplant (ASCT) in treating patients with hematologic cancer or solid tumors. Giving high-dose chemotherapy with or without TBI before ASCT stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood or bone marrow and stored. More chemotherapy may be given to prepare for the stem cell transplant. The stem cells are then returned to the patient to replace the blood forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the progression free survival (PFS) distribution for Hodgkin lymphoma (HL), non-Hodgkin lymphoma (NHL) and multiple myeloma (MM) for each disease-specific high dose therapy regimen.

SECONDARY OBJECTIVES:

I. Estimate the PFS distribution for amyloidosis, acute leukemia and selected solid tumors for each disease-specific high dose therapy regimen.

II. Explore the role of risk factors in the outcome of all treated patients. III. Examine the high dose therapy regimen-related toxicity (RRT) and overall survival after bone marrow transplant (BMT).

OUTLINE:

Patients are assigned to conditioning regimens based on disease, age, and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant hematologic disorders, amyloidosis or solid tumor malignancy
* Recurrent or refractory disease or disease at high risk for recurrence
* Hodgkin Disease (HL): Relapsed or refractory disease after chemotherapy with a minimum of one standard regimen
* Non-Hodgkin Lymphoma (NHL): (Low, Intermediate or High Grade) Relapsed or refractory disease after chemotherapy with at least one standard regimen or first complete remission (CR) lymphoblastic or small, non-cleaved cell lymphoma at high risk of relapse by high International Prognostic Index (IPI) Score
* Acute Myeloid Leukemia (AML): Low or High Risk disease in first or second CR or greater in patients in whom the risks of an allogeneic transplant outweigh the benefits
* Acute Lymphoblastic Leukemia (ALL): Low or high risk disease in first or second CR in whom the risks of an allogeneic transplant outweigh the benefits
* Multiple Myeloma (MM): Low or high risk in first or greater response (stable disease or better) or for responding patients at first progression
* Other Malignant Lymphoproliferative Disorders: (chronic lymphocytic lymphoma [CLL], Waldenstroms macroglobulinemia, relapsed or refractory disease after first-line chemotherapy
* Amyloidosis: primary or previously treated
* Solid Tumors: Testicular cancer patients who have relapsed disease or primary progressive disease which is responding to salvage therapy; relapsed or advanced-stage newly diagnosed neuroblastoma (NBL) or small round blue cell tumors (SRBCT) in patients 30 years of age; other patients with solid tumors who have recurred following conventional treatment or are at high risk for relapse, and demonstrate chemosensitivity
* Patients with malignancies who would be treated with an autologous stem cell transplant but have a syngeneic donor; a syngeneic donor would be considered to have the same risk as an autologous stem cell transplant patient
* Performance status 0-2 (Karnofsky performance status [KPS] >= 70%); patients with amyloidosis or MM with decreased KPS due to disease are eligible
* Life expectancy > 2 months
* Pulmonary function tests; diffusing capacity of the lung for carbon monoxide (DLCO) or diffusing volume of the alveolar volume (DLVA) >= 50% predicted; DLCO to be corrected for hemoglobin and/or alveolar ventilation
* Cardiac ventricular ejection fraction >= 50% by radionuclide ventriculogram or echocardiogram
* Bilirubin < 3 x normal
* Alkaline phosphatase, serum glutamic oxaloacetic transaminase (SGOT) < 3 x normal
* Calculated creatinine clearance < 40 cc/min by the modified Cockcroft-Gault formula for adults or the Schwartz formula for pediatrics
* Glomerular filtration rate by renal scan for neuroblastoma patients, to determine dosing parameters
* Positive cytomegalovirus (CMV) immunoglobulin M (IgM) and/or positive hepatitis serologies demonstrating infection will require an Infectious Disease consult and subsequent clearance
* Any active infection will require an Infectious Disease consult and subsequent clearance
* Peripheral Blood Counts of polymorphonuclear neutrophil (PMN) > 1500/uL
* Platelet (Plt) > 75,000/uL
* Prior to stem cell storage:

  * No radiation within three weeks before stem cell harvest
  * Bone marrow may be used in conjunction with blood progenitor cells
* Hematologic Malignancy patients with human immunodeficiency virus (HIV) positivity but on appropriate anti-retroviral therapy may go autotransplant with the following laboratory tests; (CD4+ cell count > 75 cells per microliter and HIV copy number < 100,000 per microliter and with Infectious Disease clearance
* Acute Leukemia, HL, NHL, MM and Solid Tumor patients must have received 2 cycles of chemotherapy followed by disease-specific restaging prior to mobilization and collection of stem cells; small round blue cell tumor patients must have received either standard therapy or surgical intervention; the disease status and response to therapy must be known prior to transplant to establish the disease status at transplant; amyloidosis patients may proceed to BMT without receiving chemotherapy
* No serious organ dysfunction unless it is caused by the underlying disease, exclusion criteria include the following:

  * Uncontrolled or severe cardiovascular disease, including recent (< 6 months) myocardial infarction, congestive heart failure, symptomatic angina, life-threatening arrhythmia or hypertension
  * Active bacterial, viral, or fungal infection
  * Active peptic ulcer disease
  * Uncontrolled diabetes mellitus
* No serious medical or psychiatric illness
* Not pregnant
* No psychiatric conditions which would prevent delivery of care; psychology clearance is necessary
* Allogeneic BMT not possible, or not desirable

  * Age > 65 years
  * No compatible donor identified
  * Estimated risk of graft vs. host disease complications greater than risk of recurrence after autologous BMT
* Adequate bone marrow or blood stem cell dose obtained:

  * For blood stem cells: total CD 34+ >= 2 x 10^6/kg or if unable to collect this dose, a total nucleated cell bone marrow dose of >= l x 10^8/kg

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2006-06-29 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip McCarthy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Leukemia: Patients diagnosed with and treated for acute myeloid leukemia or acute lymphoblastic leukemia
- Hodgkin Lymphoma: Patients diagnosed with and treated for Hodgkin Lymphoma
- Non-Hodgkin Lymphoma: Patients diagnosed with and treated for Non-Hodgkin Lymphoma
- MM/Amyloid: Patients diagnosed with or treated for multiple myeloma or amyloidosis
- Solid Tumors: Patients diagnosed with and treated for a solid tumor
Period: Overall Study
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
Started | 6 | 21 | 71 | 65 | 11
Completed | 6 | 21 | 71 | 65 | 11
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients enrolled on study and stratified by disease group as defined in statistical analysis section of protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors | Total
Number analyzed (Participants) | 6 | 21 | 71 | 65 | 11 | 174
Age, Customized [Count of Participants; unit: Participants]
  0-39 years | 1 | 8 | 6 | 3 | 9 | 27
  40-59 years | 1 | 7 | 43 | 26 | 2 | 79
  60-75 years | 4 | 6 | 22 | 36 | 0 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 23 | 29 | 3 | 71
  Male | 1 | 10 | 48 | 36 | 8 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 20 | 70 | 65 | 11 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 8 | 1 | 15
  White | 4 | 20 | 68 | 57 | 10 | 159
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 21 | 71 | 65 | 11 | 174
Risk Group [Count of Participants; unit: Participants]
  High | 6 | 10 | 43 | 10 | 11 | 80
  Standard | 0 | 11 | 24 | 44 | 0 | 79
  Unknown | 0 | 0 | 4 | 11 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Distribution of Patients With HL, NHL, and MM for Each Disease-specific High-dose Therapy Regimen, Estimate Provided for 10-yr PFS (Median Follow-up Time in Survivors)
Description: Assessed using the product-limit based Kaplan Meier method. Additionally, a 95% confidence interval of the distribution will be computed.
Time Frame: From the date of transplantation to the date of first observed disease progression or death due to any cause, assessed up to 12 years
Population: Each disease strata presents PFS for each conditioning regimen defined in the protocol
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
Number analyzed (Participants) | 6 | 21 | 71 | 65 | 11
Proportion of participants
  BuCy: number analyzed (Participants) | 6 | 7 | 27 | 0 | 0
  BuCy | 33 [0 to 71] | 14 [0 to 40] | 22 [7 to 38] |  |
  CBV: number analyzed (Participants) | 0 | 14 | 43 | 0 | 0
  CBV |  | 43 [17 to 69] | 37 [23 to 52] |  |
  VCp: number analyzed (Participants) | 0 | 0 | 1 | 0 | 7
  VCp |  |  | 0 [0 to 0] |  | 43 [6 to 80]
  Mel120: number analyzed (Participants) | 0 | 0 | 0 | 18 | 0
  Mel120 |  |  |  | 22 [2 to 41] |
  Mel200: number analyzed (Participants) | 0 | 0 | 0 | 47 | 0
  Mel200 |  |  |  | 13 [3 to 22] |
  CyTtCp: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  CyTtCp |  |  |  |  | 0 [0 to 0]
  TtC1500: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  TtC1500 |  |  |  |  | 50 [0 to 100]

2. Secondary Outcome: Regimen-related Toxicity Grade 2-4 in Any Organ (Measured by Bearman Score, Values Range From 0 (None) to 4 (Fatal))
Description: Toxicities will be reported using descriptive statistics.
Time Frame: Up to 100 days after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
Number analyzed (Participants) | 6 | 21 | 71 | 65 | 11
Participants | 1 | 9 | 19 | 31 | 3

3. Secondary Outcome: Response Rate (Complete Remission)
Description: Response rates will be reported using descriptive statistics.
Time Frame: At 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
Number analyzed (Participants) | 6 | 21 | 71 | 65 | 11
Participants | 5 | 17 | 54 | 17 | 7

4. Secondary Outcome: Overall Survival, Presented as the Estimate at 10-yrs (Median Follow-up Time in Survivors)
Description: Assessed using the product-limit based Kaplan Meier method.
Time Frame: Patients are followed up to maximum of 12 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
Number analyzed (Participants) | 6 | 21 | 71 | 65 | 11
Proportion of participants | 33 [0 to 71] | 61 [40 to 82] | 45 [33 to 57] | 39 [27 to 51] | 46 [16 to 75]

ADVERSE EVENTS:
Time Frame: SAE= 100 days after transplantation All cause mortality = 12 years
Description: SAE= Regimen related toxicity grade 2-4 in any organ system (Bearman Score, range from 0 (none) to 4 (fatal)
Arm/Group | Acute Leukemia | Hodgkin Lymphoma | Non-Hodgkin Lymphoma | MM/Amyloid | Solid Tumors
All-Cause Mortality (participants affected / at risk) | 4/6 | 8/21 | 41/71 | 45/65 | 6/11
Serious Adverse Events (participants affected / at risk) | 1/6 | 9/21 | 19/71 | 31/65 | 3/11
Other Adverse Events (participants affected / at risk) | 0/6 | 0/21 | 0/71 | 0/65 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Leukemia (N=6) | Hodgkin Lymphoma (N=21) | Non-Hodgkin Lymphoma (N=71) | MM/Amyloid (N=65) | Solid Tumors (N=11)
Regimen Related Toxicity (General disorders) | 1 (1) | 9 (9) | 19 (19) | 31 (31) | 3 (3) — Any organ system (cardiac, renal, pulmonary, lower GI, CNS, hepatic, stomatitis, bladder)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT00536601/Prot_SAP_000.pdf